CLINICAL TRIAL: NCT04132635
Title: A Randomized, Open-label, Multicenter Clinical Trial to Evaluate the Combination Efficacy of Double-layer Artificial Dermis and Growth Factor in the Treatment of Chronic Wounds Ulcer
Brief Title: A Trial to Evaluate the Combination Efficacy of Artificial Dermis and Growth Factor in Chronic Wounds Ulcer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QK-MP-201903
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Chronic Wound
MeSH Terms: interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artificial dermis with growth factor (Experimental)
  Interventions: Device: artificial dermis; Other: growth factor
- artificial dermis only (Experimental)
  Interventions: Device: artificial dermis

INTERVENTIONS:
Device: artificial dermis — artificial dermis will be used after fully debridement of the wound
Other: growth factor — growth factor
  Arms: artificial dermis with growth factor

SUMMARY:
Double layer artificial dermis repair material has been widely used in scar plastic, burn, trauma, chronic wounds and other aspects of wound repair and reconstruction. In the course of clinical application, we found that for chronic wounds, the combination of artificial dermis and growth factor can shorten the wound healing cycle, and have a positive impact on the economy and psychology of patients. In order to verify this effect, we plan to carry out this study to evaluate whether double-layer artificial dermis repair material combined with growth factor treatment can improve wound closure rate and shorten closure cycle compared with single artificial dermis for chronic wound.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as chronic wounds ulcer;
2. The affected limb has sufficient blood perfusion. The ankle brachial index was 0.65-1.3, or the partial pressure of oxygen was more than 40 mmHg, or Doppler ultrasound showed enough blood flow.
3. After debridement, the distance between the wound and the edge of other ulcers was >2cm.
4. After debridement, the area of exposed bone or tendon was >4cm2.
5. The wound was completely debridement without obvious necrosis, infection control or osteomyelitis control.
6. The duration of ulcer wound was at least 30 days.
7. Sign the informed consent voluntarily.

Exclusion Criteria:

1. Poor control of diabetes (fasting blood glucose ≥ 8.0mmol/l, HbA1c ≥ 12%);
2. The researchers think that there are factors affecting wound healing, such as the use of corticosteroids, immunosuppressants and other drugs, chemotherapy or radiotherapy within one year.
3. To receive or plan to receive drugs or treatment, the researchers believe that these drugs or treatment will interfere with or affect the speed and quality of wound healing;
4. Unstable Charcot's foot or Charcot's joint disease with bone protrusion;
5. Patients with severe lymphedema, coagulation disorders, autoimmune diseases, cardiovascular and cerebrovascular diseases, and severe hepatopulmonary and renal diseases;
6. Those who have received hyperbaric oxygen treatment within 5 days before enrollment, or who have received or plan to receive growth factor, tissue-engineered skin or other skin substitutes treatment within 30 days;
7. Those who have participated in or are participating in other clinical studies within 30 days before screening;
8. Pregnant, or lactating women;
9. Poor general condition or other conditions not suitable for the use of double-layer artificial leather repair materials;
10. Be allergic to collagen or chondroitin sulfate;
11. Other cases that researchers think are not suitable for the participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
average closure time | From the beginning of the treatment period to the time when the survival rate of skin grafting reaches 100% or 12 weeks visit (whichever comes first), record the average time when all the subjects who reach the complete closure of the wound

SECONDARY OUTCOMES:
total wound closure rate | From the beginning of the treatment period to the survival rate of skin grafting reaching 100% or 12 weeks visit (whichever comes first), record the total number of patients who have reached the complete closure of the wound during this period
  The total wound closure rate = (the number of patients who achieved complete wound closure within 12 weeks / the total number of patients in the group) * 100%.

IPD SHARING:
Plan to Share IPD: Undecided